CLINICAL TRIAL: NCT04847388
Title: Prevalence of Substance Abuse Among Anti-retroviral Treatment Naive Patients Positive for HIV Antibodies- A Cohort Study
Brief Title: Prevalence of Substance Abuse Among Anti-retroviral Treatment Naive Patients Positive for HIV Antibodies
Status: Completed | Type: Observational
Sponsor: Singh, Ranjan Kumar, M.D. (Individual)
Responsible Party: Principal Investigator, Ranjan Kumar Singh, Dr, Singh, Ranjan Kumar, M.D.
Other Study IDs: SinghRK2
Record Dates: First submitted 2021-04-11; First posted 2021-04-19 (Actual); Last update posted 2022-03-17 (Actual); Status verified 2022-03

CONDITIONS: HIV Infections
Keywords: CD4 T cell; HIV; Substance abuse
MeSH Terms: conditions — HIV Infections; Substance-Related Disorders | interventions — Ethanol; nabiximols

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- ART-naive HIV Patients with substance abuse and without substance abuse: Group A Group B
  Interventions: Drug: Substance like alcohol, marijuana, etc.
- Group A and B: Group A: ART-naive HIV seropositive with H/O substance abuse Group B: ART-naive HIV seropositive without H/O substance abuse
  Interventions: Drug: Substance like alcohol, marijuana, etc.

INTERVENTIONS:
Drug: Substance like alcohol, marijuana, etc. — Cohort study
  Other Names: Cannabis

SUMMARY:
Individuals utilise substances to elevate their mood. Alcohol, cannabis, nicotine, cocaine, and methamphetamine are examples of substances. Excessive usage of a drug that is harmful to oneself and society is referred to as substance addiction/abuse. People who inject drugs and share needles, as well as drugs that impair judgement and lead to unprotected intercourse with an infected partner, have been related to risky sex behaviour and unsafe sex, both of which increase the risk of HIV infection. Several factors, including immunologic and virologic conditions affecting host susceptibility, underlying comorbidities among drug users, use of antiretroviral therapy, and viral strain, as well as pharmacodynamic aspects of drug use, such as the pattern and type of drug administration and the route of administration, may mediate the relationship between drug use and HIV disease progression. Exacerbation of HIV progression has been shown in patients with substance addiction in laboratory research.

DETAILED DESCRIPTION:
Study of substance abuse among treatment naïve HIV patients

Background: People take substances to improve their mood. Alcohol, cannabis, nicotine, cocaine, and methamphetamine are examples of substances. Excessive usage of a drug that is harmful to oneself and society is referred to as substance addiction/abuse. These medicines have been associated to risky sex behaviour and unsafe sex, increasing the likelihood of obtaining HIV infection in two ways. People inject drugs and share needles, and drugs impair judgement, resulting in unprotected intercourse with an infected partner.

The relationship between drug use and HIV disease progression may be mediated by several factors, including immunologic and virologic conditions affecting host susceptibility, underlying comorbidities among drug users, use of antiretroviral therapy, and viral strain, as well as pharmacodynamic aspects of drug use, such as the pattern and type of drug administration and the route of administration. Laboratory based studies show exacerbation of HIV progression among patient with drug addiction.

Aim and objectives:

1. Study of prevalence of substance abuse among anti-retroviral treatment naïve patients positive for HIV antibodies.
2. To compare opportunistic infections prevalent in patients positive for HIV antibodies with substance addiction and without substance addiction.
3. To compare CD4+ T cell counts at the first visit to ART centre in patients positive for HIV antibodies with substance addiction and without substance addiction. Methods- Inclusion criteria-

1. Anti-retroviral therapy naïve patients 2. Age > 12 years Exclusion criteria-

1. 'Transferred in' patients
2. Age < 12 years. A prospective cohort studies. At Anti-retroviral therapy centre, Sadar Hospital Khagaria.

Flow chart- First visit of HIV seropositive patient-----History/clinical examination of patients H/o substance abuse (nature of substance. ? drug dependence/abuse)-------search of opportunistic infections-----------CD4 T cell count-----anti-retroviral drugs and treatment of OI, if present------follow up biweekly (first month)-----then monthly follow up for six months------CD4+ T cell count.

ELIGIBILITY:
Inclusion Criteria:

* 1. Anti-retroviral therapy naïve patients

Exclusion Criteria:

* 1. 'Transferred in' patients

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Treatment naive HIV seropositive patients
Sampling Method: Non-Probability Sample
Enrollment: 210 (Actual)
Dates: Start 2021-04-01 (Actual); Primary Completion 2022-03-15 (Actual); Study Completion 2022-03-15 (Actual)

PRIMARY OUTCOMES:
Prevalence of substance abuse among anti-retroviral treatment naïve patients positive for HIV antibodies. | One year
  Calculate prevalence (%) dividing no. of HIV patients with substance abuse by total no. of enrolled HIV patient multiplied by 100.

SECONDARY OUTCOMES:
CD4+ T cell counts at the first visit to ART centre in patients positive for HIV antibodies with substance addiction and without substance addiction. | One year
  Compare mean/SD of CD4+ T cell counts (cells/mm^3) of HIV patients in both groups at first visit to the centre by applying chi-square test.
Opportunistic infections | One year
  Comparing prevalence of opportunistic infections in both groups i.e. patients of HIV with substance abuse and Patients of HIV without substance abuse

CONTACTS AND LOCATIONS:
Overall Officials: Ranjan K Singh, Principal Investigator — Consultant Physician
Locations (1):
- ART centre, Sadar Hospital, Khagaria, Bihar, India

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kapadia F, Vlahov D, Donahoe RM, Friedland G. The role of substance abuse in HIV disease progression: reconciling differences from laboratory and epidemiologic investigations. Clin Infect Dis. 2005 Oct 1;41(7):1027-34. doi: 10.1086/433175. Epub 2005 Aug 22. PMID 16142670
- [Background] Walker HK, Hall WD, Hurst JW, editors. Clinical Methods: The History, Physical, and Laboratory Examinations. 3rd edition. Boston: Butterworths; 1990. Available from http://www.ncbi.nlm.nih.gov/books/NBK201/ PMID 21250045
- [Background] NIDA. 2019, July 29. Drug Use and Viral Infections (HIV, Hepatitis) DrugFacts. Retrieved from https://www.drugabuse.gov/publications/drugfacts/drug-use-viral-infections-hiv-hepatitis on 2021, April 5